CLINICAL TRIAL: NCT02209337
Title: Demonstrate the Safety and Preformance of the SRS Device for the Treatment of Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lyra Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-14-005
Record Dates: First submitted 2014-08-03; First posted 2014-08-05 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Anterior Vaginal Wall Prolapse; Vaginal Apex/Uterine Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SRS-I (Experimental): Implantation of SRS-I
  Interventions: Device: SRS

INTERVENTIONS:
Device: SRS

SUMMARY:
A prospective, single arm, pre-market, multi-center clinical study to evaluate the safety and performance of the SRS (Lyra Medical) vaginal mesh in POP patients

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent form and is willing to participate in the clinical study and data collection.
2. Patient age is between 18 and 75 years old
3. POP-Q: Aa and/or Ba is at least -1

Exclusion Criteria:

1. Patient is pregnant or breastfeeding
2. Patient suffering from active infection (on antibiotic therapy)
3. Patient planning vaginal delivery
4. Patient had Previous vaginal mesh surgery
5. Patient is in high risk for surgery (evidence of clinically significant cardiovascular, renal, hepatic or respiratory diseases).
6. Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.
7. Malignancy .
8. Known hypersensitivity to PEEK and polypropylene materials.
9. Participation in another investigational trial that has not completed the primary endpoint or interferes with study participation.
10. Tendency for hyper-scaring reaction
11. Diagnosed with mental or emotional disturbance.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
No device related serious adverse events | up to 12 month

SECONDARY OUTCOMES:
Minimal rate of device or procedure adverse events (intra and post operative Minimal rate of device or procedure adverse events (intra and post operative complications) | up to 12 months
Improvement in POP-Q: points Aa and Ba | up to 12 month
Improvement in POP-Q point C | up to 12 months
Achieving normal urinary function | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gil Levi, Dr., Principal Investigator — Mayanei HaYeshua Medical Center
Locations (3):
- University of Szeged, Szeged, Hungary
- Israel (2):
  - Mayanei HaYeshua Medical Center, Bnei Brak
  - Asaf HaRofeh Medical Center, Zrifin